CLINICAL TRIAL: NCT00493168
Title: Unrecognized Non-Q-wave Myocardial Infarction: Prevalence, Angiographic Correlation, and Prognostic Significance in Patients With Suspected Coronary Disease
Brief Title: Determination of the Prevalence and Prognostic Importance of Unrecognized Non-Q-wave Myocardial Infarction by MRI
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: 3434
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2007-06

CONDITIONS: Coronary Arteriosclerosis; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The first aim of this study is to determine how often unrecognized myocardial infarction occur in patients using a magnetic resonance imaging (MRI) technique (known as delayed enhancement MRI), as compared to the electrocardiogram. The second aim of this study is to determine the severity of coronary heart disease of the patients with unrecognized myocardial infarction. The final aim is to determine how the presence of unrecognized myocardial infarction detected by the MRI affects lifespan.

DETAILED DESCRIPTION:
Unrecognized myocardial infarction (MI) is known to constitute a substantial portion of lethal coronary heart disease. However, since the diagnosis of unrecognized MI is based on the appearance of incidental Q-waves on 12-lead electrocardiography, the syndrome of unrecognized non-Q-wave MI has not been described. Delayed-enhancement cardiovascular magnetic resonance (DE-CMR) can accurately identify non-Q-wave MI. The aims of this study are three-fold: 1. to determine the prevalence of unrecognized non-Q-wave and Q-wave MI, 2. to define predictors of unrecognized non-Q-wave MI, 3. to determine the prognostic significance of unrecognized non-Q-wave MI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected coronary artery disease referred for invasive coronary angiography

Exclusion Criteria:

* Clinical history of myocardial infarction
* Percutaneous coronary intervention
* Coronary artery bypass surgery
* Known uncured malignancy
* History of hypertrophic cardiomyopathy, myocarditis, or infiltrative heart disease
* Contraindication of magnetic resonance imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 1998-01; Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Han W Kim, MD, Principal Investigator — Duke Cardiovascular Magnetic Resonance Center; Raymond J Kim, MD, Principal Investigator — Duke Cardiovascular Magnetic Resonance Center
Locations (2):
- United States (2):
  - Northwestern University Medical School, Chicago, Illinois
  - Duke Cardiovascular Magnetic Resonance Center, Durham, North Carolina

REFERENCES:
- [Derived] Kim HW, Klem I, Shah DJ, Wu E, Meyers SN, Parker MA, Crowley AL, Bonow RO, Judd RM, Kim RJ. Unrecognized non-Q-wave myocardial infarction: prevalence and prognostic significance in patients with suspected coronary disease. PLoS Med. 2009 Apr 21;6(4):e1000057. doi: 10.1371/journal.pmed.1000057. Epub 2009 Apr 21. PMID 19381280